CLINICAL TRIAL: NCT03878043
Title: A Retrospective Analysis of Factors Influencing Readmission Rates of Acute Traumatic Subdural Hematoma in the Elderly
Brief Title: Factors Influencing Readmission Rates of Acute Traumatic Subdural Hematoma in the Elderly
Status: Completed | Type: Observational
Sponsor: Tarik Wasfie, MD (Industry)
Responsible Party: Sponsor-Investigator, Tarik Wasfie, MD, Professor, Department of Trauma Surgery, Ascension Health
Organization: Ascension Health (Industry)
Other Study IDs: GRMC 160013
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Traumatic Subdural Hematoma
Keywords: subdural hematoma; readmission; risk factors
MeSH Terms: conditions — Hematoma, Subdural | interventions — Aftercare

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients without Readmissions: Patients with TSDH who were not readmitted within a 6-month time period following their initial visit.
- Patients with Readmissions: Patients with TSDH who were readmitted within a 6-month time period following their initial visit.
  Interventions: Other: Follow-up Care

INTERVENTIONS:
Other: Follow-up Care — Follow up care provided upon readmission to patients who were diagnosed with a TSDH upon initial visit.
  Groups: Patients with Readmissions

SUMMARY:
Acute traumatic subdural hematomas (TSDH) readmission rate is high (27.8%) with an increase in morbidity and cost for the elderly. This study identifies risk factors affecting readmission rates for these patients and presents strategies to reduce it.

DETAILED DESCRIPTION:
A retrospective analysis was conducted on patients with traumatic brain injuries (ICD-9-CM codes 800.20 - 801.86, 852.00 - 853.05) admitted between 2014 and 2016 at Genesys Regional Medical Center through the trauma service. From this group, the investigators selected patients admitted with traumatic SDH, and those patients were followed over the following 6 months as regards to readmission status. Patients who were readmitted versus patients who were not readmitted were compared. The risk of readmission within 6 months of discharge for SDH was analyzed adjusting for age, prior anticoagulation use, Injury Severity Score (ISS), Glasgow Coma Scale (GCS), gender, time to readmission and co-morbid conditions which included diabetes mellitus, cardiovascular disease, renal disease, chronic obstructive pulmonary disease, and osteoporotic/orthopedic fractures using Cox Proportional Hazards Regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Traumatic Subdural Hematoma during time of study

Exclusion Criteria:

* Patients who expired.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to a Community General Hospital who were diagnosed with a Traumatic Subdural Hematoma.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Number of participants readmitted to the hospital | 6 months
  Number of patients diagnosed with TSDH who were readmitted to the hospital within a 6 month time frame

CONTACTS AND LOCATIONS:
Overall Officials: Tarik Wasfie, MD, Principal Investigator — Ascension Health
Locations (1):
- Genesys Regional Medical Center, Grand Blanc, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided